CLINICAL TRIAL: NCT01681355
Title: Open-label Study to Evaluate the Gastrointestinal Tolerance of a New Infant Formula in Healthy, Term, Asian Infants
Brief Title: Gastrointestinal Tolerance Study of a New Infant Formula
Acronym: BOOGIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BLU.1.C/A
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Infants
Keywords: Healthy, term, Asian infants; Infant formula
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): Healthy infants receiving standard cow's milk-based infant formula with added prebiotic oligosaccharides, and a modified fat blend and protein composition.
  Interventions: Other: Infant Formula

INTERVENTIONS:
Other: Infant Formula — Standard cow's milk based infant formula with added prebiotic oligosaccharides, and a modified fat blend and protein composition

SUMMARY:
This study is initiated to investigate the gastrointestinal tolerance of a new infant formula in healthy, term, Asian infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, well-nourished, term, Asian infants (gestational age ≥ 37 1/7 and ≤ 41 6/7 weeks)
* The mother had unequivocally decided not to exclusively breast-feed
* Formula fed for at least one week, receiving at least two formula feedings per day
* Birth weight appropriate for gestational age (AGA), 2500-4000g
* Written informed consent from parent(s) and/or legal guardian, aged ≥ 18 years.

Exclusion Criteria:

* Age > 17 weeks
* Infants known to have current or previous illnesses/conditions or intervention which could interfere with the study (impacting tolerance and/or growth), such as gastrointestinal malformations, chronic diarrhoea, malabsorptive syndrome, malnutrition, congenital immunodeficiency, or major surgery, as per investigator's clinical judgement
* Infants who suffered from gastroenteritis or diarrhoea in the last 4 weeks preceding study start.
* Infants who used any medication or nutritional supplements (except for vitamin supplementation to complement breastfeeding) in the 4 weeks preceding study start.
* Infants who have medical conditions for which a special diet other than standard (non hydrolysed) cow's milk-based infant formula is required (such as cow's milk allergy, soy protein allergy, fish protein allergy, egg protein allergy, lactose intolerance, galactosemia).
* Infants with any history of or current participation in any other study involving investigational or marketed products.
* Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol requirements.

Max Age: 17 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | up to Week 6
  Gastrointestinal tolerance is measured by stool consistency and gastrointestinal symptoms.

OTHER OUTCOMES:
Anthropometry | Week 3, Week 6
Use of medication and nutritional supplements | Week 1, Week 3, Week 6 and Week 8
Number, type and severity of (serious) adverse events | Week 1, Week 3, Week 6 and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Jan van der Mooren, PhD, Study Director — Danone Global Research & Innovation Center
Locations (5):
- Indonesia (2):
  - Panembahan Senopati Distric Hospital, Bantul, DIY Yogyakarta
  - Sakina Idaman Mothers and Children Hospital, Yogyakarta, DIY Yogyakarta
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Prince of Songkhla University Hospital, Hat Yai
  - Khon Kaen University Hospital, Khon Kaen